CLINICAL TRIAL: NCT02337621
Title: Evaluating Outcomes for Pectus Excavatum: Pain, Exercise, and Psychological Well-being
Brief Title: Pain, Exercise and Psychological Well-being in Pectus Excavatum
Acronym: PEP
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Lisa McMahon, MD, Attending, Phoenix Children's Hospital
Other Study IDs: #14-124
Record Dates: First submitted 2014-12-10; First posted 2015-01-13 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pectus Excavatum
Keywords: sunken chest; caved-in chest; chest deformity; sunken sternum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pectus excavatum surgical candidates: Any person who is eligible to undergo the Nuss procedure for surgical correction of pectus excavatum
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Recovery following major surgical procedures can be influenced by both physical (optimization of cardiopulmonary function, pain control, activity) and psychological factors. Physical activity recommendations for post-operative patients is difficult, in part because little is known about the short- and long-term benefits of exercise and mobility on post-operative pain and return to normal functioning.

DETAILED DESCRIPTION:
Major surgery has a drastic impact on the lives of patients and their families. Often, patients undergoing the Nuss procedure have lingering pain which can complicate recovery. Depending on the nature of the surgery and the severity of disease, this recovery period can be as short as a few days, or it can take several weeks and even months. Few studies have demonstrated the benefit of physical activity and exercise postoperatively on returning to normal function. Additionally, research has suggested that pain and recovery can be influenced by psychological factors.

The investigators will use wireless activity monitors to assess the activity levels of children who undergo major musculoskeletal surgery, specifically the Nuss procedure. The investigators will also evaluate this population for psychological well-being. In this pilot study, the investigators identify goals and objectives which will provide preliminary evidence for physical and psychological recommendations to reduce post-operative pain and improve recovery.

Families will be asked to complete questionnaires at different phases in the surgery (pre-surgery, post bar insertion, post bar removal). Children will be instructed to record any pain they are experiencing as a result of their condition or the surgery at various time points. The activity levels will also be followed over the course of the recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 12-18 years that are scheduled to undergo a surgical procedure for the correction of pectus excavatum

Exclusion Criteria:

* History of chronic pain disorders
* History of major mental illness such as psychosis or bipolar disorder
* Cognitive impairment significantly below average age and/or grade level
* Non-English speaking parent or child
* Unable to obtain and keep access to a cellular phone
* Loss of wireless electronic activity monitor and refusal to replace to remain in the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who are scheduled to undergo surgical correction for pectus excavatum (Nuss procedure)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Improvement in pain scores | change from baseline (2 weeks prior to bar insertion) to post bar removal surgery (3 years, 3 months)
  pain diary and self report via questionnaires
Increase in activity level/exercise | change from baseline (2 weeks prior to bar insertion) to post bar removal surgery (3 years, 3 months)
  wireless activity monitor and physical therapy notes

SECONDARY OUTCOMES:
mood | change from baseline (2 weeks prior to bar insertion) to post bar removal surgery (3 years, 3 months)
  child self report and parental report via questionnaires
body image | change from baseline (2 weeks prior to bar insertion) to post bar removal surgery (3 years, 3 months)
  child self report and parental report via modified Y-BOCS ; increased scores mean worse body image

OTHER OUTCOMES:
health related quality of life | change of quality of life from baseline (2 weeks prior to bar insertion) to post bar removal surgery (3 years, 3 months)
  child self report and parental report via PedsQL; increased scores mean better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McMahon, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fonkalsrud EW. Current management of pectus excavatum. World J Surg. 2003 May;27(5):502-8. doi: 10.1007/s00268-003-7025-5. Epub 2003 Apr 28. PMID 12715210
- [Background] Jaroszewski D, Notrica D, McMahon L, Steidley DE, Deschamps C. Current management of pectus excavatum: a review and update of therapy and treatment recommendations. J Am Board Fam Med. 2010 Mar-Apr;23(2):230-9. doi: 10.3122/jabfm.2010.02.090234. PMID 20207934
- [Background] Maagaard M, Tang M, Ringgaard S, Nielsen HH, Frokiaer J, Haubuf M, Pilegaard HK, Hjortdal VE. Normalized cardiopulmonary exercise function in patients with pectus excavatum three years after operation. Ann Thorac Surg. 2013 Jul;96(1):272-8. doi: 10.1016/j.athoracsur.2013.03.034. Epub 2013 May 14. PMID 23684487
- [Background] Tang M, Nielsen HH, Lesbo M, Frokiaer J, Maagaard M, Pilegaard HK, Hjortdal VE. Improved cardiopulmonary exercise function after modified Nuss operation for pectus excavatum. Eur J Cardiothorac Surg. 2012 May;41(5):1063-7. doi: 10.1093/ejcts/ezr170. Epub 2011 Dec 21. PMID 22219453
- [Background] Kelly RE Jr, Mellins RB, Shamberger RC, Mitchell KK, Lawson ML, Oldham KT, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Cooper D, Bagley T, Quinn A, Moskowitz AB, Paulson JF. Multicenter study of pectus excavatum, final report: complications, static/exercise pulmonary function, and anatomic outcomes. J Am Coll Surg. 2013 Dec;217(6):1080-9. doi: 10.1016/j.jamcollsurg.2013.06.019. PMID 24246622
- [Background] Nuss D, Kelly RE Jr, Croitoru DP, Katz ME. A 10-year review of a minimally invasive technique for the correction of pectus excavatum. J Pediatr Surg. 1998 Apr;33(4):545-52. doi: 10.1016/s0022-3468(98)90314-1. PMID 9574749
- [Background] Khan RS, Skapinakis P, Ahmed K, Stefanou DC, Ashrafian H, Darzi A, Athanasiou T. The association between preoperative pain catastrophizing and postoperative pain intensity in cardiac surgery patients. Pain Med. 2012 Jun;13(6):820-7. doi: 10.1111/j.1526-4637.2012.01386.x. Epub 2012 May 8. PMID 22568812
- [Background] Kelly RE Jr, Cash TF, Shamberger RC, Mitchell KK, Mellins RB, Lawson ML, Oldham K, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Bagley T, Quinn A, Moskowitz AB. Surgical repair of pectus excavatum markedly improves body image and perceived ability for physical activity: multicenter study. Pediatrics. 2008 Dec;122(6):1218-22. doi: 10.1542/peds.2007-2723. PMID 19047237
- See also: Pectus Excavatum Mobility and Stretching Exercises — https://www.youtube.com/watch?v=hy8C__bCJXM